CLINICAL TRIAL: NCT01830062
Title: Atherosclerotic Coronary Vulnerable Plaque: Correlation With Coronary Artery Calcium
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CACS NIRS
Record Dates: First submitted 2013-04-08; First posted 2013-04-12 (Estimated); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CACS and NIRS (Experimental): All patients will undergo NIRS to at least 2 major epicardial vessels as a research related intervention. Patients will be considered to be enrolled in the trial upon completion NIRS evaluation. Patients who had a clinically indicated CT with CACS evaluation within 3 months prior to the cardiac catheterization with NIRS evaluation will not have any other research related interventions. Patients who have not had a clinically indicated CT with CACS within 3 months prior to the cardiac catheterization with NIRS evaluation will have the CACS after NIRS imaging prior to discharge from the hospital.
  Interventions: Other: NIRS; Other: CACS

INTERVENTIONS:
Other: NIRS — Near infrared spectroscopy of at least 2 major epicardial vessels
  Other Names: LipiScan Coronary Imaging System, InfraReDx, Inc.
Other: CACS — Coronary artery calcium score assessed by multi-slice computed tomography

SUMMARY:
The aim of this study is to compare the relationship between the coronary artery calcification assessed by MDCT with the plaque characteristics and necrotic lipid core content of non-intervened coronary segments assessed with near infrared spectroscopy (NIRS) in patients with symptomatic coronary artery disease (CAD).

DETAILED DESCRIPTION:
A total of 60 patients, from a single center, who meet all of the study inclusion criteria and none of the study exclusion criteria will be prospectively enrolled in this study. Qualifying patients will be referred to the study site for clinically indicated, non-emergent cardiac catheterization with NIRS evaluation, either proceeded or followed by coronary artery calcium score (CACS) evaluation.

Qualifying patients that are referred directly to cardiac catheterization with NIRS assessment secondary to symptoms or abnormal functional test will be sent for cardiac CACS assessment following the catheterization before discharge from the hospital. In this group, patients who require ad hoc PCI upon initial angiography will be excluded to avoid artifacts on CACS. In patients who are referred for a clinically indicated cardiac catheterization with IVUS evaluation within 3 months after MDCT with CACS, NIRS of at least two (2) major epicardial vessels will be completed prior to any (if necessary) coronary revascularization.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥18 years of age
* Patient is clinically indicated due to angina, abnormal functional test or other ischemic symptoms to undergo non-emergent cardiac catheterization with IVUS evaluation i.If the patient has not had a cardiac MDCT with CACS meeting the protocol requirements within 3 months prior to the cardiac catheterization, the patient is able to undergo CACS following LipiScan IVUS and NIRS evaluation, prior to any coronary revascularization ii. If the patient has had a cardiac MDCT evaluation with CACS meeting the protocol requirements within 3 months prior to the cardiac catheterization, LipiScan IVUS and NIRS imaging will be completed in at least two (2) major epicardial vessels prior to any coronary revascularization
* At least two (2) major epicardial native vessels are suitable for interrogation by LipiScan IVUS imaging and NIRS evaluation, defined as:

  i.At least 30 mm of vessel that is > 2.0mm in diameter ii.No other contraindications to imaging
* No contraindications for LipiScan IVUS and NIRS evaluation
* No contraindications for CACS evaluation by MDCT
* Subject must be able to provide informed consent form and comply with the protocol requirements

Exclusion Criteria:

* Evidence of clinical hemodynamic instability in the 6 hours before either procedure
* Prior history of percutaneous coronary intervention (PCI) with stent placement
* Prior history of bypass grafts
* Female subject that is pregnant or lactating
* Any other factor that the investigator feels would put the patient at increased risk or otherwise make the patient unsuitable for participation in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Correlation between CACS and LCBI | maximum duration of 3 months between CACS and NIRS
  The primary endpoint for this study is individual patient level correlation between the total CACS of the entire coronary tree with the max LCBI4mm within the vessels imaged.

SECONDARY OUTCOMES:
Vessel level correlation of CACS and LCBI | maximum of 3 months between CACS and NIRS
  Vessel level and individual coronary artery level (LM, LAD, LCx, RCA) analysis of CACS with max LCBI4mm and total LCBI for the vessel imaged
Vessel level comparison of angiographic and IVUS parameters | maximum of 3 months between CACS and NIRS
  Vessel level comparison of angiographic and IVUS parameters with yellow plaque defined by LCBI (both max LCBI4mm and total vessel LCBI)
Segment level analysis of CACS, IVUS and lipid core plaque in patients with abnormal CT | maximum of 3 months between CACS and NIRS
  In subset of patient where coronary angiography and NIRS is driven by patient with abnormal CT coronary angiogram, the CT angiographic parameters are utilized for Segment level analysis between the CACS, IVUS and lipid core plaque

CONTACTS AND LOCATIONS:
Overall Officials: Ron Waksman, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States